CLINICAL TRIAL: NCT04711265
Title: A Longitudinal Cohort Study to Assess Sustained Immunogenicity up to 48 Months to Quadrivalent Human Papillomavirus Vaccine Among HIV-infected Girls and Boys Age 10-15 Years in Kenya
Brief Title: Antibody Response to Prophylactic QHPV Vaccine at 48 Months Among HIV-infected Girls and Boys
Status: Completed | Type: Observational
Sponsor: Kenya Medical Research Institute (Other)
Collaborators: University of Washington (Other); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Nelly Rwamba Mugo, Senior Principal Clinical Research Scientist, Kenya Medical Research Institute
Other Study IDs: KENYAMRI
Record Dates: First submitted 2020-12-08; First posted 2021-01-15 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: HPV Vaccine; HPV Infection; HIV-1-infection
Keywords: HPV Vaccine, HIV infection, Adolescents, Africa
MeSH Terms: conditions — Papillomavirus Infections; HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples for HPV antibody titer assessment HIV viral load CD4 cell count
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Quadrivalent HPV [Type 6, 11, 16 and 18] L1 Virus-Like Particle Vaccine — Intramuscular injection with 3 doses of QHPV
  Other Names: QHPV vaccine

SUMMARY:
Longitudinal observational cohort study and extension of the MISP ID: 38406 'immunogenicity and safety of quadrivalent human papillomavirus vaccine in HIV-infected pre-adolescent girls and boys in Kenya'.

DETAILED DESCRIPTION:
We evaluated for persistence of HPV antibody by measuring titers to specific HPV types 6, 11, 16 and 18 at re-enrollment month 24 , 36 and 48 months in addition to month 7 and 12, after initial vaccination. This provided data for immunogenicity among HIV-infected children for approximately 48 months after initial vaccination. We assessed decline over study intervals in HPV type-specific antibodies.

ELIGIBILITY:
Inclusion Criteria:

* receipt of 3 doses of QHPV vaccine
* participated in primary immunogenicity study
* consent/assent with parental consent for participants age <18 years
* willing to continue extended follow up for 36 months

Exclusion Criteria:

* decline consent

Ages: 9 Years to 14 Years | Sex: All
Age Groups: Child
Study Population: HIV-1 infected boys and girls who had received 3 doses of QHPV vaccine
Sampling Method: Non-Probability Sample
Enrollment: 176 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Human Papillomavirus Antibody Titers | 48 months
  Geometric mean titers for HPV type -6, -11, -16 and -18

SECONDARY OUTCOMES:
HIV RNA viral load | 48 months
  Impact of HIV RNA viral load on HPV antibody response
CD 4 cell count | 48 months
  Impact of immune status on HPV antibody response

CONTACTS AND LOCATIONS:
Locations (1):
- Partners in Health Research and Development, Thika, Kiambu County, Kenya

IPD SHARING:
Plan to Share IPD: No